CLINICAL TRIAL: NCT04501575
Title: A Feasibility Study of a Randomized Controlled Trial to Assess the Efficacy of the Osteopathic Consultation on Neck-shoulder Pain in Computer Users
Brief Title: Feasibility of RCT on the Efficacy of the Osteopathic Consultation in Computer Users
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Universidade do Porto (Other)
Responsible Party: Principal Investigator, Rui José Gomes de Pinho Santiago, PhD Student, Universidade do Porto
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: UPorto_DemSSO_RS
Record Dates: First submitted 2020-07-29; First posted 2020-08-06 (Actual); Last update posted 2020-08-06 (Actual); Status verified 2020-08

CONDITIONS: Trapezius Muscle Strain

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Osteopathic consultation (Experimental): It consists of 1 session. Each osteopathic session is based on a structural evaluation and treatment tailored to the participant-specific complains
  Interventions: Other: Osteopathic Consultation
- Osteopathic sham consultation (Sham Comparator): Osteopathic Sham treatment was applied using manual contact on specific bony surfaces using very light pressure. The practitioner was counting the seconds up to 1 minute between the areas where to apply the light touch without any intention to treat or diagnose.
  Interventions: Other: Sham Osteopathic Consultation
- Usual Care (No Intervention): Participants will be on a waiting list, and meanwhile, they are advised to deal with their pain in the way they would, but without using any sort of Manual Therapy.

INTERVENTIONS:
Other: Osteopathic Consultation — A consultation including case history taking, physical assessment, osteopathic manual treatment, exercise prescription, and postural advice.
  Arms: Osteopathic consultation
Other: Sham Osteopathic Consultation — A sham treatment using light touch on bony structures, no diagnosis, advise or prescriptions
  Arms: Osteopathic sham consultation

SUMMARY:
This study investigates the feasibility of conducting a large scale Randomized Controlled Trial (RCT) to analyze the efficacy of the osteopathic consultation in reducing the intensity of pain and changing electromyographic activity in the musculature of the neck-shoulder region for the computer user's population.

ELIGIBILITY:
Inclusion Criteria:

* Uses computer for over five hours daily, for over one year
* Reports non-specific pain over the neck-shoulder region

Exclusion Criteria:

* No neurologic signs or symptoms
* No known pathology that could mask the reported pain
* No knowledge or experience with osteopathy

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 30 (Actual)
Dates: Start 2019-09-17 (Actual); Primary Completion 2020-02-12 (Actual); Study Completion 2020-02-20 (Actual)

PRIMARY OUTCOMES:
Differences in electrical activity during typing task using surface electromyography | baseline and after 2-4 days of the treatment
  Surface electromyography (sEMG) was used to retrieve the electrical activity of the Upper Trapezius (UT) muscles. The electrical signal was normalized through the maximum isometric voluntary contraction (MIVC) and expressed as a percentage of MIVC. sEMG data will be collect at 4 different moments of the 15 minutes typing task. Electrodes placement, data collection and processing was performed according to SENIAM standards.
Differences in Pressure-pain Threshold (PPT) | baseline and after 2-4 days of the treatment
  A Digital Pressure Algometer (Wagner FORCE ONE FDIX 50', Wagner Instruments, Greenwich, CT, USA) was used on the trapezius muscle, superior fibers, both sides. The exact location on the muscles was defined as 2cm above the medial electrode, on the muscle fiber direction. During the collection of the PPT, the participant stopped the typing task and rested arms on the legs. The algometer pointer was placed perpendicular to the points marked for evaluation, and then, vertical compression force was applied. That force was increased continuously at a rate of 1 kg/cm2 until pain was reported. Measurements were made in the seating position, immediately before and after the writing task. To ensure the maximum reading was obtained, the C-Peak option of the device was enabled. Participants were instructed of the procedures in advance, and simulation on their forearm was performed before the data collection.
Difference in the self-reported intensity of pain using the numerical rating scale (NRS) | baseline, after 2-4 days of the treatment and after 1 week of the treatment
  This numeric scale, is used on its 11-point version. NRS represents a simple, 1-dimensional measuring instrument for the assessment of pain intensity (0 = no pain, 10 = unbearable pain). Participants were asked to visualize the quantity of pain they were experiencing at that precise moment over the shoulder-neck region, both sides.

SECONDARY OUTCOMES:
Satisfaction Level with the experience | 1 week after data collection for all participants.
  This questionnaire aims at retrieving satisfaction levels with the recruitment and data collection processes. It was adapted from the one used by Pflugeisen et al., (2016).

CONTACTS AND LOCATIONS:
Overall Officials: José Torres da Costa, Professor, Principal Investigator — Professor
Locations (1):
- Labiomep, Porto, Portugal

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Santiago RJ, Esteves JE, Baptista JS, Magalhaes A, Costa JT. Results of a feasibility randomised controlled trial of osteopathy on neck-shoulder pain in computer users. Complement Ther Clin Pract. 2022 Feb;46:101507. doi: 10.1016/j.ctcp.2021.101507. Epub 2021 Nov 3. PMID 34753085